CLINICAL TRIAL: NCT06695104
Title: YMCA Produce Prescription Project (YPRx)
Acronym: YPRx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tessa Mork (Other)
Collaborators: AmeriGroup (Unknown); Hungry Harvest (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); Elevance Health (Industry)
Responsible Party: Sponsor-Investigator, Tessa Mork, Association Director of Community Health, YMCA of Metropolitan Washington
Organization: YMCA of Metropolitan Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00022594; 2022-70424-38459 (Other Grant/Funding Number: USDA GusNIP award number)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pre-diabetes
Keywords: diabetes prevention program; produce rx program; produce prescription
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two study arms: intervention or control. All participants, regardless of study arm, will be enrolled in a year-long Produce Rx Program through which they will receive weekly deliveries of grocery bags containing fresh produce. Additionally, participants assigned to the intervention arm will be enrolled in a Diabetes Prevention Program, coordinated by the Y, through which they will receive health education, coaching, and peer support for a year via 26 virtual group sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Produce Rx Program Only (Control) (Active Comparator): YMCA Produce Prescription Program deliveries of fresh produce bags once per week for 52 weeks.
  Interventions: Behavioral: YMCA Produce Rx (YPRx) Program Only (Control)
- Produce Rx Program + Diabetes Prevention Program (Experimental): YMCA Produce Prescription Program deliveries of fresh produce bags once per week for 52 weeks plus the Diabetes Prevention Program via 26 virtual coaching and support sessions over 12 months.
  Interventions: Behavioral: YMCA Produce Rx (YPRx) Program + the Diabetes Prevention Program (DPP)

INTERVENTIONS:
Behavioral: YMCA Produce Rx (YPRx) Program Only (Control) — Participants in the control group will receive weekly, home-delivered produce bags of fresh vegetables and fruits and sized for each participants' household. Produce deliveries will be administered for 52 weeks.
  Arms: Produce Rx Program Only (Control)
Behavioral: YMCA Produce Rx (YPRx) Program + the Diabetes Prevention Program (DPP) — Participants will receive weekly, home-delivered produce bags of fresh vegetables and fruits and sized for each participants' household. Produce deliveries will be administered for 52 weeks. Additionally, participants will be registered for a free, year-long YMCA membership and enrolled in the DPP. Through the DPP, participants will receive health education, coaching, and peer support via 26 virtual group sessions over a year.
  Arms: Produce Rx Program + Diabetes Prevention Program

SUMMARY:
In this randomized control study, participants will be randomized 1:1 to either participate in the YMCA's Produce Prescription Program (YPRx) and receive weekly deliveries of fresh produce bags for their household or to receive YPRx plus participate in the Diabetes Prevention Program (DPP).

The investigators hypothesize that participants randomized to receive YPRx plus DPP will have greater weight loss, increased physical activity, improved diet quality and behaviors, increased food security, improved self-rated health assessment, decreased healthcare utilization from baseline to endline (12 months) compared to those randomized to receive YPRx produce deliveries only.

We will also collect data on process measures for implementation purposes.

DETAILED DESCRIPTION:
This study is a randomized control trial testing the impact of adding disease-specific, evidence-based health education (DPP) to produce prescriptions (YPRx) on participants' health. DPP is a 12-month diabetes prevention behavioral weight loss program developed by the Centers for Disease Control and Prevention and implemented nationwide. In this study, investigators will test whether the addition of health education, coaching, and peer support through DPP improves the effectiveness of YPRx. This trial will take place in the Washington D.C. Metropolitan Area in collaboration with the YMCA of Metropolitan Washington, a provider of DPP and YPRx, Hungry Harvest, a purveyor of produce deliveries, and Amerigroup/Elevance Health, a Medicaid managed care organization. Participants will be randomized 1:1 to either participate in YPRx only or to participate in YPRx plus the DPP. The length of the trial will be 12 months for each participant, and outcomes will be measured at baseline, 4 weeks, 3 months, 6 months, 9 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Recipient of Medicaid through Amerigroup
* Has never been diagnosed with type I or type II diabetes
* Access to laptop, computer, or phone with internet, or willing to use a provided device
* District of Columbia resident
* Available to attend DPP classes at the scheduled recurring day and time
* Not pregnant

Exclusion Criteria:

* Under the age of 18
* Not a recipient of Medicaid through Amerigroup
* Has been diagnosed with type I or type II diabetes
* No access to laptop, computer, or phone with internet
* Not a resident of the District of Columbia
* Cannot attend DPP classes at the scheduled recurring day and time
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-06 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline, 3 months, 6, months, 9 months, and 12 months
  Change in body weight will be measured by change in absolute pounds and percent of body weight. Participants will provide self-reported weight in pounds via quarterly online surveys at baseline, 3 months, 6 months, 9 months, and 12 months (endline).

SECONDARY OUTCOMES:
Change in physical activity | Baseline, 3 months, 6, months, 9 months, and 12 months
  Change in physical activity will be measured by the change in absolute minutes of physical activity and percent change in time spent being physically active. Minutes spent being physically active over the past 7 days, self-reported via quarterly online surveys at baseline, 3 months, 6 months, 9 months, and 12 months (endline).
Change in food security status | Baseline and 12 months
  Change in food insecurity will be measured using the 6-question U.S. Household Food Security Screener Module which ask participants about food security within the household framed around personal and familial food consumption based on the ability to afford food in the past 30 days. Responses will be self-reported via online surveys at baseline and endline (12 months).
Change in participant dietary intake | Baseline and 12 months
  Change in dietary intake will be measured using the National Cancer Institute's Dietary Screener Questionnaire. Frequency of food and beverage consumption over the previous month will be self-reported by participants via online surveys at baseline and endline (12 months). Foods and beverages include: "Pure Fruit Juices", "Fruit", "Green Leafy or Lettuce Salad", "Fried Potatoes", "Other Kinds of Potatoes", "Cooked Beans", "Vegetables", "Salsa", "Pizza", and "Tomato Sauce". Responses to all questions will be measured using 11-point scale ranging from "Never" to "6 or more times per day" for "Pure Fruit Juices", a 9-point scale ranging from "Never" to "2 or more times per day" for all other food categories, plus an additional response option "Don't know/Prefer not to answer" for each question.
Change in participant food behaviors | Baseline and 12 months
  Change in food behavior will be measured as the change in number of days (0-7) the participant, or someone else in their family, cooked dinner at home during the preceding week. Frequencies will be self-reported by participants via online surveys at baseline and endline (12 months).
Change in personal health self-rated health assessment | Baseline and 12 months
  Change in self-rated health assessment will be measured by the change in participant's self-rated health assessment collected via online survey at baseline and 12 months using a five-point Likert scale ("Poor" to "Excellent") .
Change in participant healthcare utilization- self-reported | Baseline and 12 months
  Change in healthcare utilization will be measured by the change in frequency of accessing healthcare during the three months preceding baseline and endline. This outcome will be measured by whether or not the participant accessed various types of medical attention ("Yes", "No" "Don't know/Prefer not to answer"), and if so, how many times ("None" to "16 or more" plus "Don't know/Prefer not to answer") as self-reported via online surveys at baseline and endline (12 months).

OTHER OUTCOMES:
Change in participant healthcare utilization- healthcare records | Baseline and 12 months
  Change in healthcare utilization will be measured by comparing healthcare claims data at baseline and endline (12 months).
Change in participant HbA1c | Baseline and 12 months
  Change in participant HbA1c will be measured by the absolute change and percent change in HbA1c levels retrieved from healthcare claims data at baseline and endline (12 months).
YMCA Produce Rx (YPRx) program satisfaction- quantitative process measure | 4 weeks, 3 months, 6 months, 9 months, 12 months
  Participant satisfaction with the YMCA Produce Rx program will be self-reported via online surveys at 4 weeks, 3 months, 6 months, 9 months, 12 months. Questions will include rating: the experience measured on a 6-point Likert scale ("Very negative" to "Very positive" plus "Don't know/Prefer not to answer"), the quality of produce measured on a 5-point Likert scale ("Very high quality" to "Very low quality"), familiarity with the produce measured on a 4-point Likert scale ("Very familiar, I received produce I already purchased and ate often" to "Very new, I received produce that was unfamiliar or new to me"), the quantity of produce measured on a 3-point Likert scale ("Not enough, I ran out and would have liked to have more" to "Too much, I often had leftover produce that I didn't use").
YMCA Produce Rx (YPRx) program satisfaction- qualitative process measure | 4 weeks, 3 months, 6 months, 9 months, 12 months
  Participant satisfaction with the YMCA Produce Rx program will be self-reported via online surveys. One question asks about difficulties or challenges with the program and is presented at 4 weeks, 3 months, 6 months, 9 months, and 12 months (endline). A second question asks if there is anything else the participant would like to share and is presented at 12 months only. Both questions will be measured using written responses submitted in open text boxes.
Self-perceived YMCA Produce Rx (YPRx) program impact- quantitative measure | 12 months
  Self-perceived impact of the YMCA Produce Rx program on participants will be self-reported via an online survey at endline (12 months). Four questions ask participants about the program's impact on their excitement toward learning about healthy eating, ability to eat healthier, and ability to save time and money, using a 5-point Likert scale from "Strongly Disagree" to "Strongly Agree".

CONTACTS AND LOCATIONS:
Overall Officials: Kristy McCarron, MPH, Principal Investigator — YMCA of Metropolitan Washington; Julia Wolfson, PhD MPP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- YMCA of Metropolitan Washington, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided